CLINICAL TRIAL: NCT03398629
Title: Diagnosis and Management of Intrauterine Growth Restriction, Structural Anomalies and Chromosomal Anomalies: A Prospective Cohort Study
Brief Title: Diagnosis and Management of Intrauterine Growth Restriction and Congenital Anomalies
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Wei Zhong, Director, Guangzhou Women and Children's Medical Center
Other Study IDs: 2017120501
Record Dates: First submitted 2017-12-05; First posted 2018-01-12 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Intrauterine Growth Restriction; Fetal Anomaly; Chromosomal Anomalies; Pregnancy
MeSH Terms: conditions — Fetal Growth Retardation; Congenital Abnormalities; Chromosome Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years

GROUPS / COHORTS (3):
- IUGR group: Estimated fetal weight below10th percentile for gestational age associated with Abnormal Doppler flow in the umbilical cord (umbilical artery pulsatility index (PI)>95th percentile).
- Structural anomaly group: Fetus/neonates/infants who are diagnosed as congenital malformations, deformations, disruptions, dysplasias by ultrasound.
- Chromosomal anomaly group: Fetus/neonates/infants diagnosed by genetic amniocentesis or chorionic villus sampling for increased risk for fetal aneuploidy or fluorescence in situ hybridization.

SUMMARY:
The purpose of this prospective cohort study is to build a large platform that includes clinical information (prenatal diagnosis and postnatal follow-up data) and biological specimen banks of fetuses/infants with IUGR or congenital anomalies, which provide vital support and research foundation for accurate diagnosis, precision treatment and meticulous management.

DETAILED DESCRIPTION:
Intrauterine growth restriction (IUGR) and congenital anomalies are one of the important reasons for infant and childhood death, which carry a high burden to affected individuals and their families. The detection rates are increasing with the improving diagnostic techniques. There are several cohorts mentioning the screening of these diseases during pregnancy. However, at present there have been no reported relevant cohorts that study from intrauterine to extrauterine period to understand and research the occurrence and development of IUGR and congenital anomalies as well as the relationship between IUGR and the presence of congenital anomalies. So in this study, the investigators aim to conduct large-sample prospective cohort study based on clinical data and biological samples to observe the occurrences, progression and clinical outcomes of IUGR and congenital anomalies, and investigate factors, pathogenesis and prognostic biomarkers of these diseases. These results can play an important role in preventing the occurrence of IUGR and congenital anomalies, promoting prognosis and guiding the clinical treatments.

All pregnant women or neonates/infants who present to Guangzhou Women and Children's Medical Center with the diagnoses of IUGR or congenital anomalies (including congenital malformation, deformations, disruptions, dysplasia and chromosomal anomalies) are eligible to participate in the study. Investigators will use routine obstetrical ultrasound to evaluate the growths and developments of fetuses during pregnancy. Investigators will collect dietary habits, exposures (the usage of medicine, exposure to contaminants), maternal history and history of disease, imaging data from the pregnant women who are prenatally diagnosed with fetus having IUGR or congenital anomalies. Afterbirth, the neonates will receive appropriate treatment. Regular physical and neural development examination with a pediatrician to measure growth and development that has taken place. Data regarding diagnosis, treatment, growth and development will be collected by intelligent data extraction platforms. Machine learning and statistical analysis are used to build the diagnostic prediction models to improve the accuracy of prenatal diagnosis of IUGR and congenital anomalies. In addition, the investigators will estimate the burden on individuals and families by evaluating the associations between interventions during pregnancy and after birth and clinical outcomes such as adverse events, length of hospitalization, hospitalization expenses in abnormal children.

In particular, maternal blood, placenta, cord blood, child' blood, urine, stool and tissue and other specimens during hospitalization and outpatient clinical visit will be collected and stored in the biospecimen bank. biospecimen bank is managed by special accounts to ensure the correct and ethical usage of specimens. Investigators hope to identify some markers that impact the prognosis of IUGR and congenital anomalies by analyzing the prenatal and postnatal serologic data. Genetic testing will be done on some fetuses to help identify the pathogenesis and the most appropriate treatment.

ELIGIBILITY:
Inclusion Criteria:

All pregnant women who present to Guangzhou Women and Children's Medical Center meeting one of the following prenatal diagnoses and neonates/infants who are diagnosed as one of the following anomalies will be invited to participate:

1. Intrauterine growth restriction (IUGR)
2. Structural anomaly
3. Chromosomal anomaly

Exclusion Criteria:

1. Pregnant women who don't agree to participate;
2. Pregnant women delivering babies at other hospitals.
3. Prenatally suspected anomalies that are not confirmed by postnatal diagnosis.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population includes pregnant women present to Guangzhou Women and Children's Medical Center with prenatal diagnosis of IUGR, congenital malformations, deformations, disruptions, dysplasia or chromosomal anomalies; and neonates/infants with conformed IUGR, congenital malformations, deformations, disruptions, dysplasia or chromosomal anomalies.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2038-03-01 (Estimated); Study Completion 2038-03-01 (Estimated)

PRIMARY OUTCOMES:
Consistency between prenatal and postnatal diagnosis of fetal anomalies | At delivery
  Comparison of results of prenatal ultrasound or genetic amniocentesis and results of postnatal diagnosis in neonates with anomalies.
Constituent ratio of all types of anomalies among live infants | At delivery
  Including constituent ratio of all types of anomalies in prenatal diagnosis and constituent ratio of anomalies confirmed by clinical diagnosis after births.
Differences of mortality rates between infants with prenatal diagnosis and those with postnatal diagnosis | up to 1 year
Differences of Kaup's indexes between IUGR infants with prenatal intervention and those with postnatal intervention | up to 1 year
  Kaup's index＝weight(kg)÷height(cm)^2×10^4
Recovery of organ functions following postnatal management in infants with anomalies | up to 5 years

SECONDARY OUTCOMES:
Catch-up growth for weight | up to 2 years
  Weight was measured in infants at 4, 6, 9, 12, 15, 18, 21 and 24 months after birth.
Catch-up growth for height | up to 2 years
  Height was measured in infants at 4, 6, 9, 12, 15, 18, 21 and 24 months after birth.
Neurodevelopment at childhood | at age of 1 year old]
  Including adaptive, gross motor, fine motor, language and personal-social, assessed by Gesell Developmental Schedules.
Intelligence quotient | At age of 6 years
  Assessed using Wechsler's Intelligence Scale for Children-Ⅳ(WISC-Ⅳ) consisting of verbal test and performance test. Verbal test covers the following areas: information, vocabulary, arithmetic, comprehension and similarities; Performance test includes picture completion, picture arrangement, block design, object assembly and coding. Each subscale scores range: 1 to 19. Higher scores indicate better performance. A total score is computed by summing the 10 subscale scores. Full-scale intelligence quotients is calculated based on the Wechsler's Intelligence Scale for Children-Ⅳ total score according to instructions. It ranges from 40 to 160, in which under 70 is defined as mental retardation.
Quality of life | At age of 5-12 years
  Assessed using Pediatric Quality of Life Inventory including physical, emotional, social and school scales. Total Scale score = 23 items, Physical Health Summary Score = 8 items, Psychosocial Health Summary Score = 15 items. Each question is answered on the "5-point Likert scale from 0 (never) to 4 (almost always)". Then "items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. The mean of the scores on the 100-point scale is then calculated (sum of all items divided by number of items answered). The total score ranges from 0 to 100, and higher scores indicate a better quality of life.
Parental psychological distress after a prenatal or postnatal diagnosis of anomaly. | up to 42 days postpartum
  Parental psychological distress was assessed by using Brief Symptom Inventory (53-item-self-report instrument) which consists of nine subscales: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobia, paranoia and psychoticism. Respondents rank each feeling item on a 5-point scale ranging from 0 (not at all) to 4 (extremely). The subscale and total scores are calculated as an average of the relevant items, with higher scores indicating more severe psychopathology. The test scores are reported in terms of standardized area T-scores.
Parental quality of life after a prenatal or postnatal diagnosis of anomaly. | up to 42 days postpartum
  Parental quality of life was assessed by using World Health Organization Quality of Life Scale Brief which consists of four subscales: physical health with 7 items, psychological with 6 items, social relationships with 3 items and environment with 8 items. Each item is rated on a 5-point Likert scale. Each item is scored from 1 to 5 on a response scale. Raw domain scores were transformed to a 4-20 score according to guidelines. The mean score of items within each domain is used to calculate the domain score. After computing the scores, they transformed linearly to a 0-100-scale. A higher score indicates higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhong, Master, Principal Investigator — Guangzhou Women and Children's Medical Center
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided